CLINICAL TRIAL: NCT00005058
Title: A Direct Comparison of Contrast Enhanced Power Doppler Ultrasound in Primary Breast Cancer and Axillary Nodal Status With Histopathological Variables and Clinical Outcome
Brief Title: Enhanced Ultrasound in Determining Extent of Disease in Women With Primary Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000067655; RMNHS-1443; EU-20003
Record Dates: First submitted 2000-04-06; First posted 2004-04-12 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2005-04

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — High-Energy Shock Waves

INTERVENTIONS:
Procedure: ultrasound imaging

SUMMARY:
RATIONALE: New imaging procedures, such as enhanced ultrasound may improve the ability to determine the extent of breast cancer.

PURPOSE: Diagnostic study of enhanced ultrasound in women who have locally advanced primary breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Measure blood flow of primary breast lesions and corresponding lymph nodes by Power Doppler Ultrasound (PDU) and compare this information with metastatic potential and patient survival in women with primary breast cancer. II. Correlate intratumor/-nodal blood flow with pathological variables using standard histology and special stains in this patient population. III. Correlate intratumor microvessel density with total tumor blood flow and with the presence of axillary lymph node metastases using this diagnostic method in these patients. IV. Correlate tumor blood flow with various markers of angiogenesis using this diagnostic method in these patients. V. Compare tumor blood flow as measured with PDU before and after contrast enhancement in these patients.

OUTLINE: This is a diagnostic study. Patients receive ultrasound contrast agent IV. An ultrasound probe with Power Doppler facility is swept over the skin surface in a standard fashion before and after contrast enhancement. Blood flow data is acquired over the volume of the mass and/or lymph nodes using a video recorder. The scanning time ranges between 5 to 15 minutes depending on the size and exact location of the breast mass and axillary lymph nodes. Within 1 week of the ultrasound, patients undergo surgery and the mass and axillary lymph nodes are removed.

PROJECTED ACCRUAL: Approximately 200 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Clinically suspected locally advanced breast cancer where treatment indicated is primary surgery (wide local excision or simple mastectomy) and axillary dissection (clearance) Inflammatory breast cancer eligible No recurrent disease Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No New York Heart Association class III or IV heart disease At least 14 days since prior myocardial infarction Pulmonary: No severe chronic obstructive pulmonary disease Other: No galactosemia No mental illness or handicap

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior neoadjuvant chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics At least 1 month since prior core biopsy (Tru-cut) of breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-08

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gui, MD, MS, FRCS(Edin), FRCS(Eng), Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Trust, London, England, United Kingdom